CLINICAL TRIAL: NCT01437891
Title: An Open-label Clinical Outcomes Study to Determine the Safety and Efficacy of Sentra AM® and Sentra PM® for Post-traumatic Stress Disorder and Gulf War Fibromyalgia
Brief Title: Sentra AM® and Sentra PM® for Post-traumatic Stress Disorder (PTSD) and Gulf War Fibromyalgia (GWF)
Acronym: GWF001
Status: Completed | Type: Observational
Sponsor: Stephanie Pavlik (Industry)
Responsible Party: Sponsor-Investigator, Stephanie Pavlik, Clinical Research Associate, Targeted Medical Pharma
Organization: Targeted Medical Pharma (Industry)
Other Study IDs: GWF001
Record Dates: First submitted 2011-09-15; First posted 2011-09-21 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Post-traumatic Stress Disorder; Persian Gulf Syndrome
Keywords: PTSD; Military veteran; Gulf War; Fibromyalgia; Gulf War Syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Persian Gulf Syndrome; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An open-label clinical outcomes study to determine the safety and efficacy of Sentra AM® and Sentra PM® for post-traumatic stress disorder (PTSD) and Gulf War fibromyalgia (GWF).

DETAILED DESCRIPTION:
Male and female military veterans age 18 to 75 experiencing moderate to severe PTSD symptoms including cognitive dysfunction, sleep disorders and mood disorders.

Open-label internet questionnaire-based clinical outcomes study. 250 subjects. 60 days from enrollment initiation to completion and study close. Sentra AM- two capsules given orally once daily in the morning for 30 days. Sentra PM- two capsules given orally once daily thirty minutes before bedtime for 30 days.

To measure improvement in quality of life determined by the change in short form-36 (SF-36) general health survey.

Improvements in daytime sleepiness determined by the Epworth Sleepiness Scale (ESS), improvement in cognitive and emotional function using the Cognitive emotion regulation questionnaire - short (CERQ-Short), change in PTSD symptoms with the Primary Care - PTSD (PC-PTSD), Psychopathy Checklist- Military (PCL-M). Heart rate variability (HRV) data variation will be measured in a group of twenty subjects.

ELIGIBILITY:
Inclusion Criteria:

1. United States military veterans reporting PTSD and/or Gulf War Illness symptoms at least three months after return from duty.
2. Men and non-pregnant, non-lactating women over the age of 18 and under the age of 75, able to read and understand English-language informed consent.
3. Men and women of child-bearing potential willing to use adequate contraception, not to become pregnant or impregnate their partner for the study duration.
4. Patients who will continue on a stable dose (no less than three months) of other medications they are taking and maintain the same dose throughout the duration of the study.
5. Patients willing to commit to completing all clinical questionnaires and guidelines during study-related procedures.

Exclusion Criteria:

1. Patients who have previously taken Sentra AM or Sentra PM.
2. Patients not fluent in English.
3. Participation in a clinical trial within one (1) month prior to screening.
4. Uncontrolled or unstable serious cardiovascular, pulmonary, gastrointestinal, endocrine or neurologic disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female military veterans age 18 to 75 experiencing moderate to severe PTSD symptoms including cognitive dysfunction, sleep disorders and mood disorders.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
SF-36 general health survey | Baseline and Day 30
  A general health questionnaire to measure quality of life. Change from baseline.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | Baseline and Day 30
  Improvements in daytime sleepiness determined by the Epworth Sleepiness Scale.
CERQ-short | Baseline and Day 30
  Assessment of cognitive function. Change from baseline.
PCL-Military | Baseline and Day 30
  Changes in symptoms of military specific PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: William Shell, MD, Principal Investigator — Targeted Medical Pharma, Inc.
Locations (1):
- Targeted Medical Pharma, Los Angeles, California, United States